CLINICAL TRIAL: NCT01052623
Title: Status of the Growth Hormone/ Insulin-like Growth Factor-1 (GH/IGF-1) Axis in Relation to Growth Failure, Body Weight and Neuroprotection in Children With Ataxia Telangiectasia
Brief Title: Status of Growth Hormone/ Insulin-like Growth Factor-1 (GH/IGF-1) Axis and Growth Failure in Ataxia Telangiectasia (AT)
Acronym: GHAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Dr. Stefan Zielen, Johann Wolfgang Goethe University Hospitals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FRA.GHAT.2009
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Ataxia Telangiectasia; Growth Failure
Keywords: GH/IGF-1; Ataxia telangiectasia (AT); IGF-1 Generation Test; Growth hormone
MeSH Terms: conditions — Ataxia Telangiectasia; Failure to Thrive | interventions — Human Growth Hormone; Clonidine; Estradiol; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Growth hormone-testing (GH/IGF-1-testing) (Experimental): Patients (girls over 8 years and boys over 10 years) are primed with estradiol 1 mg orally for 2 days, to help avoid false results of growth hormone (GH) levels in blood samples. Then provocation testing is done, with two tests back to back. It determines blood levels of GH and the body's response to testing with drugs called arginine and clonidine. Patients are admitted to the pediatric inpatient unit and will have an intravenous (IV) line placed in the arm. Arginine is given by IV over 30 minutes, and blood samples are taken as indicated.
  The next day, the clonidine test is performed according to current guidelines. Then the IGF-1 generation test is done to see if the patient has the ability to generate IGF-1 in response to injections of GH for 5 consecutive days.
  Interventions: Drug: Somatropin, Clonidine, L-Arginin-Hydrochloride, Estradiol valerate

INTERVENTIONS:
Drug: Somatropin, Clonidine, L-Arginin-Hydrochloride, Estradiol valerate — 1 mg Estradiol valerate with for two days before GH-testing pre pubertal girls older than 8 years and pre pubertal boys older than 10 years. L-Arginin-Hydrochloride in the vein (0.5 g/kg KG maximum dose 30g) over 30 minutes. Clonidine orally (0,075 mg/m2 BSA). Somatropin-NutropinAq subcutaneum,a single one shot (dose 0.03 mg/KG, daily, over five days).
  Other Names: Catapressan; Growth hormone; NutropinAq; Progynova 21 mite; L-Arginin_hydrochlorid-einmolar

SUMMARY:
This study will evaluate the status of the growth hormone/ insulin-like growth factor-1 (GH/IGF-1) axis in relation to growth failure, body weight and composition and neuroprotection in children with Ataxia telangiectasia (AT).

DETAILED DESCRIPTION:
Growth failure and GH/IgF-1 deficiency has been described in patients diagnosed with Ataxia telangiectasia (AT) [Boder et al.,1958]. This condition is a fatal inherited disease caused by a mutation of the ATM gene on chromosome 11 leading to chromosomal instability, immunodeficiency, cancer susceptibility and and endocrinological abnormalities. In this regard, several groups demonstrated a cross-linking of ATM with growth factor pathways. Participation of the ATM protein in insulin signaling through phosphorylation of eIF-4E-binding protein 1 has been postulated [Yang et al.,2000]. Peretz et al.[2001] described that expression of the insulin-like growth factor-I receptor is (IGF-I R) ATM dependent in a pathway regulating radiation response. In addition, Shahrabani-Gargir et al.[2004] found that the ATM gene controls IGF-I R gene expression in a DNA damage response pathway. Suzuki et al.[2004] described that IGF-I phosphorylates AMPK-alpha, a key regulator of cholesterol and fatty acid synthesis, acts in an ATM-dependent manner . We have recently demonstrated reduced levels of circulating Insulin-like growth factor-I (IGF-I) and its main binding protein 3 (IGFBP-3) in AT patients accompanied with decreased body mass index [Schubert et al.,2005]. Furthermore, apart from regulating somatic growth and metabolism, evidence suggests that the GH/IGF-I axis is involved in the regulation of brain growth, development and myelination. Moreover, GH and particularly IGF-1 have potential neuroprotective effects in different in vitro and in vivo experimental models. In addition we have recently shown that extracerebellar MRI-lesions in AT go along with deficiency of the GH/IGF-1 Axis, markedly reduced body weight, high ataxia scores and advanced age [Kieslich et al.,2009]. Supplementation with these growth hormones might overcome the progressive dystrophy and may have clinical benefits against the progression of neurodegeneration and immunodeficiency.

We found that supplementation with GH significantly increased longevity of Atm-deficient mice and improve T-cell immunity and locomotor behaviour [Schubert et al.,2009]. Surprisingly IGF-1 was not generated in the ATM deficient mice, indicating that the GH/IGF-1 signalling is impaired. Taken this into account a accurate diagnostic approach of the GH/IGF-1 axis is mandatory including a IGF-1 generation test before long term treatment either with GH or IGF-1 is justified in humans.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of AT
* Have no fusion of epiphyses/closed growth plates as determined by X-ray of left wrist and hand (special skeletal age film)
* Be between 3 years to 18 years old and have not completed puberty
* Consent to permit blood and/or tissue samples for storage
* Demonstrate growth failure: height below the 10th percentile for chronological age
* Have a primary care physician at home
* Demonstrate growth failure, defined as growth velocity (measured as linear growth) that is less than 5% to 10% of that expected for children of the same age group, over the past 12 months
* Willingness to remain hospitalized for several days
* Provide evidence of serum IGF-1 level performed within the preceding 6 months and the results fall below 25% range of normal limits for age

Exclusion Criteria:

* Have fusion of epiphyseal plates
* Be under the age of 3 years or have reached completion of puberty
* Have a serum IGF-1 level that is above the 25% range of normal limits for age
* Be above the 10th percentile height for chronological age
* Demonstrate any history of anaphylactic reaction or hypersensitivity to one of the GH formulation
* Have any active or suspected neoplasia
* Demonstrate signs of intracranial hypertension as evidenced by papilledema upon examination by fundoscopy
* Have any condition that, in the investigator's opinion, places the patient at undue risk by participating in the study
* Be unwilling to undergo testing or procedures associated with this protocol
* Have acute or chronic infections
* Have a hypersensitivity to one of the drugs: Clonidine hydrochlorid, Arginine hydrochlorid, Estradiol valerate, Somatropin
* Have a presence of bradycardia, cardiac arrhythmia, have symptoms of a sick sinus syndrome
* Suffer from depression
* Have acute or recurrent thrombosis
* Have acute liver diseases

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the GH increase after Arginine Provocation Test | at minute 0, 30, 60, 90 und 120 after infusion

SECONDARY OUTCOMES:
The GH increase after Clonidine Provocation Test. To evaluate the safety and efficacy of the IGF-1 generation test. To correlate GH/IgF-1 deficiency to BMI To correlate GH/IgF-1 deficiency to MRI findings | at minute 0, 30, 60, 90 und 120 after dosing of Clonidin. IgF-1 generation test after 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof. Dr., Principal Investigator — Children´s Hospital, Goethe-University
Locations (1):
- Children's Hospital, Goethe-University, Frankfurt am Main, Germany

REFERENCES:
- [Background] BODER E, SEDGWICK RP. Ataxia-telangiectasia; a familial syndrome of progressive cerebellar ataxia, oculocutaneous telangiectasia and frequent pulmonary infection. Pediatrics. 1958 Apr;21(4):526-54. No abstract available. PMID 13542097
- [Background] Lavin MF. Ataxia-telangiectasia: from a rare disorder to a paradigm for cell signalling and cancer. Nat Rev Mol Cell Biol. 2008 Oct;9(10):759-69. doi: 10.1038/nrm2514. PMID 18813293
- [Background] Schubert R, Reichenbach J, Zielen S. Growth factor deficiency in patients with ataxia telangiectasia. Clin Exp Immunol. 2005 Jun;140(3):517-9. doi: 10.1111/j.1365-2249.2005.02782.x. PMID 15932513
- [Background] Isgaard J, Aberg D, Nilsson M. Protective and regenerative effects of the GH/IGF-I axis on the brain. Minerva Endocrinol. 2007 Jun;32(2):103-13. PMID 17557036
- [Background] Yang DQ, Kastan MB. Participation of ATM in insulin signalling through phosphorylation of eIF-4E-binding protein 1. Nat Cell Biol. 2000 Dec;2(12):893-8. doi: 10.1038/35046542. PMID 11146653
- [Background] Peretz S, Jensen R, Baserga R, Glazer PM. ATM-dependent expression of the insulin-like growth factor-I receptor in a pathway regulating radiation response. Proc Natl Acad Sci U S A. 2001 Feb 13;98(4):1676-81. doi: 10.1073/pnas.98.4.1676. Epub 2001 Feb 6. PMID 11172010
- [Background] Shahrabani-Gargir L, Pandita TK, Werner H. Ataxia-telangiectasia mutated gene controls insulin-like growth factor I receptor gene expression in a deoxyribonucleic acid damage response pathway via mechanisms involving zinc-finger transcription factors Sp1 and WT1. Endocrinology. 2004 Dec;145(12):5679-87. doi: 10.1210/en.2004-0613. Epub 2004 Sep 2. PMID 15345673
- [Background] Suzuki A, Kusakai G, Kishimoto A, Shimojo Y, Ogura T, Lavin MF, Esumi H. IGF-1 phosphorylates AMPK-alpha subunit in ATM-dependent and LKB1-independent manner. Biochem Biophys Res Commun. 2004 Nov 19;324(3):986-92. doi: 10.1016/j.bbrc.2004.09.145. PMID 15485651
- [Background] Kieslich M, Hoche F, Reichenbach J, Weidauer S, Porto L, Vlaho S, Schubert R, Zielen S. Extracerebellar MRI-lesions in ataxia telangiectasia go along with deficiency of the GH/IGF-1 axis, markedly reduced body weight, high ataxia scores and advanced age. Cerebellum. 2010 Jun;9(2):190-7. doi: 10.1007/s12311-009-0138-0. PMID 19898915
- [Background] Schubert R, Schmitz N, Pietzner J, Tandi C, Theisen A, Dresel R, Christmann M, Zielen S. Growth hormone supplementation increased latency to tumourigenesis in Atm-deficient mice. Growth Factors. 2009 Oct;27(5):265-73. doi: 10.1080/08977190903112663. PMID 19626507
- See also: Related Info — http://www.info-at.de